CLINICAL TRIAL: NCT04725838
Title: The UPGRADE Study: Real World Outcomes® of Differential Target Multiplexed (DTM-SCS®) Stimulation in Existing and New Medtronic Implants
Brief Title: Differential Target Multiplexed Spinal Cord Stimulation (DTM-SCS®) Real World Outcomes
Status: Completed | Type: Observational
Sponsor: Celéri Health, Inc. (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: UPGRADE
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Medtronic Intellis™ and Vanta™ — Differential Target Multiplexed (DTM®) programming using Medtronic's Intellis™ or Vanta™ Spinal Cord Stimulation systems

SUMMARY:
The UPGRADE registry will capture long-term, real-world outcomes to understand the effect of Differential Target Multiplexed (DTM®) programming in the Spinal Cord Stimulation (SCS) implanted population on the management of chronic pain, primarily on its use for trunk and/or limb pain. The clinical study is sponsored by Celéri Health and is funded through a financial grant from Medtronic's External Research Program. The registry study will be conducted across approximately 25 centers in the United States with up to 600 participants enrolled.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, observational, open-label, non-randomized, multi-center study. It is designed to collect clinical follow-up data on Differential Target Multiplexed (DTM®) programming that is available in Medtronic's Intellis™ and Vanta™ spinal cord stimulators, which has shown superiority to conventional programming parameters in a randomized controlled trial (NCT03606187).

Participants currently implanted with a permanent neurostimulation system, whom are planned for conversion to DTM® programming as well as newly identified participants planned to undergo a trial of neurostimulation using DTM® will be eligible to participate in this study. Data will be collected at baseline prior to DTM® programming exposure.

Participants who continue to meet eligibility criteria and have had their implanted DTM programming activated will enter a follow-up period for up to 24 months, where participant self-reported questionnaires will be assessed each month with study visits to occur at months 12 and 24.

Throughout the study, objective functional data will be collected automatically as part of the Medtronic device interrogation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must provide written informed consent prior to any clinical study-related procedure.
2. Participant is at least 18 years (or the minimum age required by local law to consent for participation in a clinical investigation) or older at the time of enrollment.
3. Participant has a permanent Medtronic Intellis™ neurostimulation system implanted or is planning to be implanted with a Medtronic Intellis™ or Vanta™ neurostimulation system.
4. Participant has access to an iPhone or Android capable device and/or computer with regular internet access for the purposes of electronically completing web-based participant self-reported questionnaires via SMS text or email.

Exclusion Criteria:

1. Participant is unable to provide written informed consent or to comply with study-related requirements, procedures, and visits.
2. Participant is a profound responder for all pain areas to existing neurostimulation therapy (≥80% reported relief).
3. Participant is enrolled, or intends to participate, in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug, or additional testing beyond standard of care procedures) which could confound the results of this trial as determined by the investigator.
4. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the participant's ability to participate in the clinical investigation or to comply with follow-up requirements.
5. Participant is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant has a permanent Medtronic Intellis™ neurostimulation system implanted or is planning to be implanted with a Medtronic Intellis™ or Vanta™ neurostimulation system and is a candidate for Differential Target Multiplexed (DTM®) programming for the management of chronic pain, primarily on its use for trunk and/or limb pain.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the Pain Impact Score as measured by the PROMIS-29 before and after introduction of Differential Target Multiplexed (DTM®) stimulation programming in a real-world population. | 24 months

SECONDARY OUTCOMES:
To characterize the responder rate for pain by pain area per Percent Pain Relief for DTM-SCS® compared to participant baseline treatment. | 24 months
To characterize the responder rate for pain by pain area per Numeric Rating Scale for DTM-SCS® compared to participant baseline treatment. | 24 months
To evaluate the longitudinal characterization of objective posture and activity measures. | 24 months
  Time spent in each activity/position (Intellis™ device data)
To characterize Patient Global Impression of Change (PGIC) with neurostimulation. | 24 months
To evaluate the performance of the DTM® pre-programming questionnaire in predicting outcome of DTM-SCS® programming. | 24 months
To characterize the neuropathic pain quality using PROMIS-Neuropathic Pain Quality (PROMIS-PQ-Neuro) before and after treatment. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fishman, MD, Study Director — Chief Medical Officer
Locations (34):
- United States (34):
  - Neuroversion, Anchorage, Alaska
  - Desert Sky Spine & Sports Medicine, Oro Valley, Arizona
  - Desert Sky Spine & Sports Medicine, Sierra Vista, Arizona
  - NuVation Pain Group - Buena Park, Buena Park, California
  - NuVation Pain Group - Los Angeles, Los Angeles, California
  - Spine and Sports Specialty Medical Group, Orange, California
  - Spine & Nerve Diagnostic Center - Roseville, Roseville, California
  - Florida Pain Medicine - Brandon, Brandon, Florida
  - Jax Spine & Pain Centers - Fleming Island, Fleming Island, Florida
  - Jax Spine & Pain Centers - UF North, Jacksonville, Florida
  - Jax Spine & Pain Centers - Jacksonville, Jacksonville, Florida
  - Florida Spine & Pain Specialists, Riverview, Florida
  - Jax Spine & Pain Centers -St. Augustine, Saint Augustine, Florida
  - Florida Pain Medicine - Wesley Chapel, Wesley Chapel, Florida
  - National Spine and Pain Centers - Winter Park, FL, Winter Park, Florida
  - Centurion Spine & Pain Centers (Jax Spine), Waycross, Georgia
  - Millennium Pain Center (National Spine and Pain Centers - Bloomington, IL), Bloomington, Illinois
  - National Spine and Pain Centers - National Harbor (Oxon Hill), Oxon Hill, Maryland
  - National Spine and Pain Centers - Pikesville, MD, Pikesville, Maryland
  - Comprehensive and Interventional Pain Management, Henderson, Nevada
  - National Spine and Pain Centers - The Pain Management Center - Voorhees, Voorhees Township, New Jersey
  - Carolinas Research Institute - Mallard Creek, Charlotte, North Carolina
  - Carolinas Research Institute - Huntersville, Huntersville, North Carolina
  - Premier Pain Treatment Institute - Hillsboro, Hillsboro, Ohio
  - Premier Pain Treatment Institute - Loveland, Loveland, Ohio
  - Premier Pain Treatment Institute - Mt. Orab, Mount Orab, Ohio
  - Oklahoma Pain Physicians - Norman, Norman, Oklahoma
  - Oklahoma Pain Physicians - Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Pain Physicians - Purcell, Purcell, Oklahoma
  - North Texas Orthopedics & Spine Center- Keller/Alliance, Fort Worth, Texas
  - North Texas Orthopedics & Spine Center - Grapevine, Grapevine, Texas
  - Precision Spine Care, Tyler, Texas
  - Valley Pain Consultants, Winchester, Virginia
  - Northwest Pain Care, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — https://celerihealth.com/